CLINICAL TRIAL: NCT01158599
Title: An Open-label, Uncontrolled Phase 4 Study to Assess the Safety and Immunogenicity of the Japanese Encephalitis (JE) Vaccine Ixiaro® (IC51) in an Elderly Population
Brief Title: This is a Study to Assess the Safety and Immunogenicity of Ixiaro® (IC51) in an Elderly Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IC51-315
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Japanese Encephalitis
Keywords: Japanese Encephalitis; Vaccination; Ixiaro; elderly population
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IXIARO 0,5 ml (Other): IXIARO®, 0.5 ml (6 µg), intramuscular (i.m.) injection, two vaccinations, Days 0 and 28
  Interventions: Biological: IXIARO®

INTERVENTIONS:
Biological: IXIARO® — IXIARO®, 0.5 ml (6 µg), intramuscular (i.m.) injection, two vaccinations, Days 0 and 28

SUMMARY:
This is an open-label, uncontrolled phase 4 study to assess the safety and immunogenicity of the Japanese encephalitis (JE) vaccine Ixiaro® (IC51) in an elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 65 years of age at the time of 1st vaccination of good general health status including subjects with pharmacologically controlled conditions like hypercholesterolemia, hypertension, cardiovascular disease or non insulin-dependent diabetes mellitus
* Weight: ≥ 45.5 kg and ≤ 150 kg at Visit 0 (Screening Visit)
* White blood cells ≥2,500/mm3 and <11,000/mm3 at Visit 0
* Absolute neutrophil count within normal limits at Visit 0
* Platelets within normal limits at Visit 0
* Written informed consent obtained from the subject prior to any study related procedures

Exclusion Criteria:

* History of clinical manifestation of any flavivirus infection (Yellow Fever, Dengue Fever, JE, Tick Borne Encephalitis (TBE) and West Nile Fever/Neuroinvasive Disease)
* Vaccination against JE (including study participation in any previous or current IC51/IXIARO® clinical study), Yellow fever, Dengue Fever or West Nile Fever at any time prior or during the study
* Vaccination against TBE within 30 days prior to first IXIARO® vaccination at Visit 1 (Day 0) and until Visit 3 (Day 70)
* Use of any other investigational or non-registered medicinal product within 30 days prior to IXIARO® vaccination at Visit 1 (Day 0) and throughout the entire study period
* Immunodeficiency including status post-organ-transplantation or immuno-suppressive therapy, and a family history of congenital or hereditary immunodeficiency
* Infection with the human immunodeficiency virus (HIV, a negative test result within 30 days before screening is acceptable), Hepatitis B virus (HBV, Hepatitis B surface antigen [HBsAg]) or Hepatitis C virus (HCV)
* Administration of chronic (defined as longer than 14 days) immunosuppressants or other immune-modifying drugs within 30 days prior to IXIARO® vaccination at Visit 1 (Day 0) and during the study until Visit 3 (Day 70). (For corticosteroids this means prednisone or equivalent >= 0.05 mg/kg/day; topical and inhaled steroids are allowed).
* Periodic steroid injections, e.g., intra-articular, are not allowed within 30 days prior to first IXIARO® vaccination at Visit 1 (Day 0) and until Visit 3 (Day 70)
* History of autoimmune disease, including Type I Diabetes mellitus. Subjects with vitiligo or thyroid disease taking thyroid hormone replacement are not excluded.
* Acute febrile infections or exacerbation of chronic infection on the day of IXIARO® vaccination (Day 0 and Day 28)
* Skin cancer in the past six months. If treatment for skin cancer was successfully completed more than six months ago and the malignancy is considered to be cured, the subject may be enrolled. Subjects with history of skin cancer must not be vaccinated at the previous site of the malignancy.
* Any other malignancy in the past 5 years. If treatment for cancer was successfully completed more than 5 years ago and the malignancy is considered to be cured, the subject may be enrolled.
* Clinically significant hematological, renal, hepatic, pulmonary, central nervous, cardiovascular or gastrointestinal disorders, which are not adequately controlled by medical treatment within the last 12 weeks before IXIARO® vaccination at Visit 1 (Day 0) as judged by the site's Principal Investigator
* Clinically significant mental disorder not adequately controlled by medical treatment
* History of Guillain-Barré-Syndrome (GBS).
* History of severe hypersensitivity reactions, in particular to a component of the IXIARO® vaccine (e.g. protamine sulfate), anaphylaxis or severe cases of atopy requiring emergency treatment or hospital admission
* History of urticaria after hymenoptera envenomation, drugs, physical or other provocations, or of idiopathic cause
* Drug addiction within 6 months prior to Visit 0 and throughout the entire study period (including alcohol dependence, i.e. more than approximately 60 g alcohol per day, or conditions which might interfere with the study conduct)
* Inability or unwillingness to avoid more than the usual intake of alcohol (> 60 g alcohol/day) during the 48 hours after each vaccination
* Any condition which might interfere with study objectives or would limit the subject's ability to complete the study in the opinion of the investigator
* Persons who are committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities) will not participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Rate of subjects with serious adverse events (SAEs) and medically attended adverse events (AEs) during the vaccination period and until Day 70 after the first vaccination | until day 70

SECONDARY OUTCOMES:
Rate of subjects with SAEs and medically attended AEs during the vaccination period and up to 6 months after the second vaccination | up to 6 months
Rate of subjects with unsolicited AEs up to Day 70 after the first vaccination | up to Day 70
Rate of subjects with unsolicited AEs up to six months after the second vaccination | up to 6 months
Rate of subjects with abnormal safety laboratory parameters (hematology, clinical chemistry, urinalysis) up to Day 70 after the first vaccination | up to Day 70
Rate of subjects with solicited local and solicited systemic AEs assessed with a subject diary for 7 consecutive days after each vaccination | 7 consecutive days after each vaccination
GMTs and SCRs for JEV neutralizing antibodies determined by PRNT at Day 70 | Day 70

CONTACTS AND LOCATIONS:
Locations (5):
- Austria (2):
  - Institut für Spezifische Prophylaxe und Tropenmedizin, Vienna, Vienna
  - Medical University of Vienna - Klinische Pharmakologie, Vienna, Vienna
- Germany (3):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg
  - Universitätsklinikum Rostock, Rostock, Rostock
  - Berliner Centrum Reise- und Tropenmedizin, Berlin, State of Berlin